### **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the effects of transcutaneous electrical nerve stimulation (TENS) on chemotherapy-induced peripheral neuropathy (CIPN)

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Protocol URCC-19085 "Wireless Transcutaneous electrical nerve stimulation (TENS) for chemotherapy-induced peripheral neuropathy (CIPN): A phase II clinical trial" (NCT# 04367480)

### **Overview and Key Information**

### What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have peripheral neuropathy that was caused by your chemotherapy, which is often called CIPN. Peripheral neuropathy refers to the conditions that result when nerves that carry messages to and from the brain and spinal cord from and to the rest of the body are damaged or diseased.

# Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

This study is being done to answer the following question:

• Can we decrease the symptoms of your CIPN using a wireless transcutaneous electrical nerve stimulation device, which is often called a TENS device?

Protocol Version Date: 06/25/2021 

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your CIPN. The usual approach is defined as care most people get for CIPN.

# What is the usual approach to my CIPN?

The usual approach for patients who are not in a study is treatment with drugs that help other types of neuropathic pain (nerve pain); for example, pain that occurs with diabetes. No treatments have been approved by the Food and Drug Administration (FDA) to specifically treat symptoms of CIPN.

# What are my choices if I decide not to take part in this study?

You may choose to have the usual approach described above. You may choose to take part in a different research study, if one is available.

# What will happen if I decide to take part in this study?

If you decide to take part in this study, you will either get an active wireless TENS device for up to 6 weeks or you will get a placebo wireless TENS device for up to 6 weeks. The placebo device is a device that looks the same as the active device but does not deliver the therapeutic stimulation.

No matter what group you are in, you will receive an active device for free for personal use after you complete the 6-week study period.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the device may not improve your CIPN symptoms.

There is also a risk that you could have side effects from the device.

Some of the most common side effects that the study doctors know about are:

- Skin irritation caused by wearing the device
- Abnormal sensations

There may be some risks that the study doctors do not yet know about.


#### **Benefits**

There is evidence from a small study in humans that suggests that this TENS device may be effective in reducing CIPN symptoms. It is not possible to know now if the TENS device will improve your CIPN symptoms compared to the usual approach. This study will help the study doctors learn things that will help people with CIPN in the future.

# If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide not to participate in the study, you can follow-up with your health care provider regarding your CIPN symptoms.

### Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (University of Rochester Cancer Center NCI Community Oncology Research Program (URCC NCORP) Research Base). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.


### What is the purpose of this study?

You developed CIPN during your chemotherapy. The purpose of this study is to test if a wireless TENS device can reduce your CIPN symptoms. The effects of the active wireless TENS device will be compared to a placebo wireless TENS device. The placebo device is a device that looks the same as the active device but does not deliver the therapeutic stimulation. There will be about 150 people taking part in this study.

# What are the study groups?

This study has 2 study groups. You will not be told which group you are in.

#### Group 1

If you are in this group, you will get the active wireless TENS device and the electrodes that stick to your skin that you need for the device to work. The device is FDA approved to treat chronic pain, but has not been approved to treat all of the symptoms that often come with CIPN (for example tingling and numbness). You will be asked to wear the device below your knee for 5 hours/day for 6 weeks. You will be asked to change the leg that you wear it on each day. There will be about 75 people in this group.

### Group 2

If you are in this group, you will get the placebo wireless TENS device and the electrodes that stick to your skin that go with the device. There will be about 75 people in this group. If you receive the placebo device during the study, you will be offered the active TENS device for free after you complete the study.

Regardless of which study group you are in, you will receive an active TENS device to keep after completion of the study, but you will have to purchase the electrodes to continue to use the device.



What exams, tests, and procedures are involved in this study?

Protocol Version Date: 06/25/2021 *URCC19085(Amd3)* 

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you may have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

- Conditioned Pain Modulation Test will be used to measure nerve activity. This test includes 2 temporary pain stimuli. One involves applying pressure to your trapezius muscle (the large muscle that extends from the back of your head and neck to your shoulder) until you first feel pain and pain. The other involves pain caused by putting your hand in cold water for between 15 seconds and 1 minute. You will be allowed to remove your hand before the 15 seconds if it becomes too painful.
- Your balance will be evaluated by testing how long you can stand with your feet in different positions.
- The ability of your feet to feel light touch will be tested with a series of small fibers.

If you choose to take part in this study, you will be asked to fill out forms with questions about your CIPN symptoms and how they have affected your life, your emotional well-being, your physical function and activity, changes that you experience during the study, and your opinion about the study device. Researchers will use this information to learn more about how well the TENS device works to treat CIPN symptoms and the parts of your life that the CIPN symptoms may interfere with.

Since these forms are being used for research, the responses you provide will not be shared with your study doctor. If you have any serious health issues or other concerns, please talk with your doctor or nurse right away.

You will be asked to fill out these forms at 2 times:

- At the time that you receive the study device
- After you have used the device for 6 weeks.

The forms will take about 20-30 minutes to complete each time. You don't have to answer any question that makes you feel uncomfortable.

You will also be asked to complete a daily diary during the  $1^{st}$ ,  $4^{th}$ , and  $6^{th}$  week of the study. The diary will ask you to rate 5 neuropathy symptoms and record whether you take certain pain medications each day. The entry should take no longer than 2 minutes / day.

You will be contacted by the coordinator 4 weeks after you finish the last study visit to ask if you are still using the TENS device.


Study staff will help you download an app on your mobile device or tablet and show you how to connect to the internet and upload your TENS data. You will upload this data once a day, which will take a few minutes / day.

# What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the study device may not improve your CIPN symptoms.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

#### Side Effect Risks

There is a risk that you could have other side effects from the study device.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Known side effects are mild. Although unlikely, it is possible that other unknown side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust how long they suggest you use the device to try to reduce side effects.

#### **Device Risks**

The list below shows the most common side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

Some of the most common side effects that the study doctors know about are:

Protocol Version Date: 06/25/2021 URCC19085(Amd3)

- Skin irritation
- Abnormal sensations. In an earlier study using TENS, of the 26 participants that received TENS, 3 experienced new abnormal sensations in their feet and legs. These new abnormal sensations went away when the participants stopped using the device.

The FDA considers TENS, which is currently approved to treat chronic pain, as having non-significant risk, which means that the agency does not require that they monitor studies that use this device because of low risk to participants.

#### **Study Procedure Risks**

You will experience temporary acute pain during the Conditioned Pain Modulation test.

# What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking for CIPN. It is not necessary to report medications and supplements you are taking for other conditions.
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study
- Complete a daily diary to rate your CIPN symptoms and indicate whether you took Tylenol or NSAIDs each day during the baseline and 4<sup>th</sup> and 6<sup>th</sup> weeks of the study.
- Be willing and able to not start any new pain medications or change dosages of any currently used pain medications during the duration of the study other than Tylenol or NSAIDs.
- Login once a day to the App that the study team installs on your mobile device or tablet while the device is connected to the internet for the 6 week study period.

**For women**: Do not get pregnant while taking part in this study. Tell your study doctor right away if you think that you have become pregnant during the study.

# What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your CIPN.

This includes:

- The costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- Your insurance co-pays and deductibles.


Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study.

#### These include:

• The conditioned pain modulation test, the balance exam, and the test to see how well your feet can feel objects.

You or your insurance provider will NOT have to pay for the TENS device while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your CIPN. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

If you do not have a cellular data plan you may have to pay a small data charge for using the study App.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

# What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?


Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as results of study tests and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

#### Some of these organizations are:

- The study sponsor, the University of Rochester Cancer Center NCI Community Oncology Research Program Research Base
- Neurometrix, the company providing the TENS devices and app to upload data.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The NCI and the groups it works with to review research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

# Where can I get more information?


You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) at (\*insert telephone number\*).


# **Contact for Future Research**

Date of signature\_\_\_\_\_

| • | • | meone on the study team earch in the future. | m, may contact me or my doctor to | o sec |
|---|---|---|---|---|
| YES | NO | | | |
| My signature a | greeing to take | part in the study | | |
| | | | discussed it with the study doctored and dated copy of this form. | and |
| Participant's sig | nature | | | |
| Date of signature | | | | |
| Signature of per | son(s) conductii | ng the informed consen | nt discussion | |
